CLINICAL TRIAL: NCT03748784
Title: An Open Label Phase 1 Study of ADVM-022 (AAV.7m8-aflibercept) in Neovascular (Wet) Age-Related Macular Degeneration
Brief Title: ADVM-022 Intravitreal Gene Therapy for Wet AMD
Acronym: OPTIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADVM-022-01
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Wet Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration
Keywords: Choroidal Neovascularizatio; ADVM-022; CNV; ADVM-022-01; AAV.7m8; Anti-VEGF therapy; Blindness; Gene therapy; Aflibercept (Eylea); Age-Related Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; AAV Vector; Adverum; wAMD; AMD; wet AMD
MeSH Terms: conditions — Blindness; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, dose-ranging clinical study to evaluate the safety and tolerability of ADVM-022 in subjects with wet AMD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): 6E11 vg of ADVM-022
  Interventions: Biological: ADVM-022
- Dose 2 (Experimental): 2E11 vg of ADVM-022
  Interventions: Biological: ADVM-022

INTERVENTIONS:
Biological: ADVM-022 — ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-deficient adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Other Names: AAV.7m8-aflibercept

SUMMARY:
ADVM-022 (AAV.7m8-aflibercept) is a gene therapy product developed for the treatment of neovascular (wet) age-related macular degeneration (wet AMD). Wet AMD is a serious condition and the leading cause of blindness in the elderly. The available therapies for treating wet AMD require life-long intravitreal (IVT) injections every 4-12 weeks to maintain efficacy. A one-time IVT administration of ADVM-022 has the potential to treat wet AMD by providing durable expression of therapeutic levels of intraocular anti-VEGF protein (aflibercept) and maintaining the vision of patients. ADVM-022 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with wet AMD receiving anti-VEGF therapy in clinical practice.

DETAILED DESCRIPTION:
This open-label, multicenter, dose-ranging study will evaluate 2 dose levels in up to 30 subjects (15 per dose) with active choroidal neovascularization (CNV) secondary to AMD. Subjects who are under active anti-VEGF treatment and have demonstrated a meaningful response to anti-VEGF therapy will be considered for participation in this study. The primary endpoint for this study is safety and tolerability of ADVM-022. All subjects will continue to be assessed for 104 weeks following treatment with ADVM-022.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* Diagnosis of neovascular (wet) AMD
* BCVA ETDRS Snellen equivalent between ≤20/32 and ≥20/320 for each cohort
* Subjects must be under active anti-VEGF treatment for wAMD and received a minimum of 2 injections within 4 months prior to screening
* Demonstrated a meaningful response to anti-VEGF therapy
* Willing and able to provide consent

Exclusion Criteria:

* History of retinal disease in the study eye other than wet AMD
* Fibrosis or atrophy, retinal epithelial tear in the center of the fovea in the study eye, or any condition preventing visual acuity improvement
* History of retinal detachment (with or without repair) in the study eye
* History of vitrectomy, trabeculectomy, or other filtration surgery in the study eye
* Uncontrolled glaucoma in the study eye
* Any prior treatment with photodynamic therapy or retinal laser for the treatment of wet AMD and any previous therapeutic radiation in the region of the study eye
* Any previous intraocular or periocular surgery on the study eye within 6 months
* Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months
* Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Type, severity, and incidence of ocular and systemic adverse events (AEs) | 104 weeks
  Type, severity, and incidence of ocular and systemic adverse events (AEs)

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) | 104 weeks
  Change in best corrected visual acuity (BCVA)
Change in central subfield thickness (CST) and macular volume measured by SD-OCT | 104 weeks
  Change in central subfield thickness (CST) and macular volume measured by SD-OCT
Percentage of subjects requiring anti-VEGF injections over time | 104 weeks
  Percentage of subjects requiring anti-VEGF injections over time
Mean number of anti-VEGF injections over time | 104 weeks
  Mean number of anti-VEGF injections over time
Percentage of subjects without intraretinal fluid over time | 104 weeks
  Percentage of subjects without intraretinal fluid over time
Percentage of subjects without subretinal fluid over time | 104 weeks
  Percentage of subjects without subretinal fluid over time

CONTACTS AND LOCATIONS:
Overall Officials: OPTIC Medical Monitor, Study Chair — Adverum Biotechnologies, Inc.
Locations (11):
- United States (11):
  - Adverum Clinical Site, Bakersfield, California
  - Adverum Clinical Site, Beverly Hills, California
  - Adverum Clinical Site, Golden, Colorado
  - Adverum Clinical Site, Deerfield Beach, Florida
  - Adverum Clinical Site, Reno, Nevada
  - Adverum Clinical Site, Philadelphia, Pennsylvania
  - Adverum Clinical Site, West Columbia, South Carolina
  - Adverum Clinical Site, Nashville, Tennessee
  - Adverum Clinical Site, Abilene, Texas
  - Adverum Clinical Site, Houston, Texas
  - Adverum Clinical Site, The Woodlands, Texas

REFERENCES:
- [Derived] Khanani AM, Boyer DS, Wykoff CC, Regillo CD, Busbee BG, Pieramici D, Danzig CJ, Joondeph BC, Major JC Jr, Turpcu A, Kiss S. Safety and efficacy of ixoberogene soroparvovec in neovascular age-related macular degeneration in the United States (OPTIC): a prospective, two-year, multicentre phase 1 study. EClinicalMedicine. 2023 Dec 22;67:102394. doi: 10.1016/j.eclinm.2023.102394. eCollection 2024 Jan. PMID 38152412